CLINICAL TRIAL: NCT05376592
Title: Association of Genomic Polymorphisms With Cancer Cachexia in Subjects With Pancreatic Adenocarcinoma
Brief Title: Assoc. of Genomic Polymorphisms With Cancer Cachexia in Subjects With Panc Adenocarcinoma
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00083490; LCI-SUPP-PDAC-CC-001 (Other: Atrium Health)
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pancreas Adenocarcinoma; Cachexia
Keywords: Cancer Cachexia; Wasting Syndrome; Pancreatic Cancer
MeSH Terms: conditions — Cachexia; Wasting Syndrome; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood or buccal sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A major complication of pancreatic adenocarcinoma (PDAC) is cancer cachexia (CC) which is a complex syndrome characterized by skeletal muscle mass loss (with or without loss of fat mass) and progressive functional impairment not reversible by conventional nutritional support. It is estimated to occur in over 75% of patients with advanced PDAC, the highest incidence of all solid tumors, and contributes significantly to poor outcomes and mortality. Though there is overlap amongst the pathophysiologic studies evaluating CC in murine models of different tumor types, the high prevalence of CC within gastrointestinal (GI) malignancies and specifically PDAC suggest that dedicated studies evaluating polymorphisms in candidate genes specific to PDAC warrant further evaluation. The collection and analysis of specimens under this study will facilitate the identification and characterization of genomic polymorphisms associated with CC in PDAC patients. Subsequently, this data may help contribute towards diagnostic and therapeutic treatments that may improve patient outcomes.

DETAILED DESCRIPTION:
This pilot study consists of a cohort of 100 locally advanced unresectable or metastatic PDAC subjects with a prospective analysis of biomarkers that may be associated with CC, a major negative prognostic factor in outcomes.

The study protocol-directed assessments consist of four experimental measures (gene single nucleotide polymorphisms and available clinical information including weights, imaging review of sarcopenia, and select labs) used to determine factors that potentially contribute to CC in subjects with PDAC. Main confounding factors to be evaluated include stage of disease, receipt of anti-cancer therapies, and sites of metastatic disease.

Specimens collected from PDAC patients treated at Atrium Health Wake Forest Baptist Comprehensive Cancer Center may include blood or buccal swabs. Specimens may be collected during any standard of care clinic visit after screening and confirmation of eligibility.

Collected and processed specimens will be stored for analysis at Atrium Health and analyzed in the Nutrition Research Institute (NRI). All specimen results will remain deidentified. Personal health information will be collected on study participants and linked to results of genomic analysis but will be deidentified prior to any data analysis and presentation at scientific conferences, sharing with non-Atrium Health investigators and for publications.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of personal health information by the subject in accordance with the practices of the Levine Cancer Institute and Atrium Health. NOTE: HIPAA authorization will be included in the informed consent.
* Male or female patients age ≥ 18 years at the time of consent
* Histological or cytological confirmation of pancreatic adenocarcinoma, with a diagnosis of locally advanced unresectable PDAC (LAPC) or metastatic pancreatic adenocarcinoma. LAPC is defined as per NCCN 16. Note: Subject can be enrolled at any time during their cancer course following histologic diagnosis.
* Able to provide a blood or buccal sample.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with pancreatic adenocarcinoma will be will be approached for potential consent during a clinic visit at any participating Levine Cancer Institute location.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Cancer cachexia (CC) | approx. 3 months
  A binary variable will be determined for each subject indicating if they have developed CC within 3 months after diagnosis as defined as weight loss of at least 5%.

SECONDARY OUTCOMES:
Cancer cachexia (CC) | approx. 3 months
  A binary variable will be determined for each subject indicating if they have developed CC within 3 months after diagnosis as defined as weight loss of at least 10%.
Sarcopenia | approx. 3 years
  A binary variable will be determined for each subject indicating if they have developed sarcopenia at any point in time of or after diagnosis. Measurements of sarcopenia will be obtained via body composition analysis of available, routine CT and/or MRI imaging.
Overall Survival (OS) | approx. 3 years
  Overall survival is defined as the duration of time from the date of diagnosis to the date of death from any cause.
One-year survival | approx. 1 year
  One-year survival will be determined as a binary variable for each subject indicating if the subject is alive one year after the date of diagnosis.
Progression free survival (PFS) | approx. 3 years
  Progression free survival is defined as the duration from date of diagnosis to first occurrence of either progressive disease or death.

CONTACTS AND LOCATIONS:
Overall Officials: Kunal Kadakia, MD, Principal Investigator — Atrium Health Levine Cancer Institute
Locations (2):
- United States (2):
  - Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No